CLINICAL TRIAL: NCT01666977
Title: A Phase 1b/2 Trial of AMG 386 in Combination With Pemetrexed and Carboplatin as First Line Treatment of Metastatic Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Phase 1b/2 Trial of AMG386 With Pemetrexed and Carboplatin in Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20101128; 2011-001111-31 (EudraCT Number)
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — trebananib; Pemetrexed; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Experimental): Arm A: AMG 386 placebo IV QW, pemetrexed 500 mg/m2 IV Q3W, carboplatin AUC 6 IV Q3W, for up to 6 cycles
  Interventions: Drug: AMG 386 Placebo; Drug: Pemetrexed; Drug: Carboplatin
- Arm B (Experimental): Arm B: AMG 386 15 mg/kg IV QW, pemetrexed 500 mg/m2 IV Q3W, carboplatin AUC 6 IV Q3W, for up to 6 cycles
  Interventions: Drug: AMG 386; Drug: Pemetrexed; Drug: Carboplatin
- Arm C (Experimental): Arm C: AMG 386 30 mg/kg IV QW, pemetrexed 500 mg/m2 IV Q3W, carboplatin AUC 6 IV Q3W, for up to 6 cycles
  Interventions: Drug: AMG 386; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: AMG 386 — 15mg/kg
  Arms: Arm B
Drug: AMG 386 — 30 mg/kg
  Arms: Arm C
Drug: AMG 386 Placebo — AMG 386 Placebo
  Arms: Arm A
Drug: Pemetrexed — Pemetrexed 500 mg/m2
Drug: Carboplatin — Carboplatin AUC 6

SUMMARY:
The purpose of this phase 1b/2 study is to estimate the treatment effect of study drug measuring progression free survival.

DETAILED DESCRIPTION:
To evaluate the incidence of adverse events and clinical laboratory abnormalities defined as dose-limiting toxicity in subjects with metastatic non-squamous non-small cell lung cancer (NSCLC) treated with AMG 386 in combination with pemetrexed and carboplatin

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable stage IV non-squamous non small cell lung cancer (NSCLC)
* Radiographically evaluable disease (measurable or non-measurable) per RECIST 1.1 with modifications
* Adequate hematological, renal, and hepatic function, normal coagulation profile, calculated CrCL ≥ 45 mL/min
* Other criteria may apply

Exclusion Criteria:

* Any prior chemotherapy or targeted therapy for non-squamous NSCLC
* Subjects with adenosquamous histology or any histology subtype containing greater than 10% squamous cells
* Subjects with an epidermal growth factor receptor (EGFR) mutation sensitive to treatment with a tyrosine kinase inhibitor (TKI)
* Subjects with known anaplastic lymphoma kinase (EML4-ALK) translocations
* History or presence of central nervous system metastases
* Central (chest) radiation therapy within 28 days prior to enrollment/randomization, radiation therapy to any other site(s) within 14 days prior to enrollment/randomization
* History of pulmonary hemorrhage or gross hemoptysis within 6 months
* History of arterial or venous thromboembolism within 12 months
* History of clinically significant bleeding within 6 months
* Clinically significant cardiovascular disease within 12 months
* Other criteria may apply

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Incidence of adverse events and clinical laboratory abnormalities defined as a DLT
  Subjects will be evaluated for progression free survival.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (35):
- United States (13):
  - Research Site, Fayetteville, Arkansas
  - Research Site, Hot Springs, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, Palm Springs, California
  - Research Site, Pleasant Hill, California
  - Research Site, San Diego, California
  - Research Site, Santa Monica, California
  - Research Site, Peoria, Illinois
  - Research Site, Paducah, Kentucky
  - Research Site, Hannover, New Hampshire
  - Research Site, The Bronx, New York
  - Research Site, Bismarck, North Dakota
  - Research Site, Greenville, South Carolina
- Australia (7):
  - Research Site, Camperdown, New South Wales
  - Research Site, Kogarah, New South Wales
  - Research Site, Randwick, New South Wales
  - Research Site, Tweed Heads, New South Wales
  - Research Site, Herston, Queensland
  - Research Site, Bentleigh East, Victoria
  - Research Site, Heidelberg, Victoria
- Research Site, Brussels, Belgium
- Canada (7):
  - Research Site, Hamilton, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
- Greece (4):
  - Research Site, Heraklion
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Spain (3):
  - Research Site, Málaga, Andalusia
  - Research Site, Zaragoza, Aragon
  - Research Site, Madrid, Madrid

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com